CLINICAL TRIAL: NCT03686436
Title: Vitreomacular Interface Abnormalities Indiabetic Retinopathy Using Ocular Coherence Tomography
Brief Title: Vitreomacular Interface Abnormalities in Diabetic Retinopathy Using OCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, seham dahy, ophthalmology specaliist, Assiut University
Other Study IDs: seham dahy
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: on Vitreomacular Interface Abnormalities in Diabetic Retinopathy
Keywords: unrecognized condition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ocular coherence tomography — imaging by ocular coherence tomography

SUMMARY:
to evaluate vitreomacular interface abnormalities in diabetic retinopathy by using Ocular Coherence Tomography (OCT)

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is a leading health concern and a major cause of blindness .DR can be complicated by scar tissue formation, macular edema tractional retinal detachment. Optical coherence tomography has found patient with DR has diffuse retinal thickening , cystoid macular edema ,posterior hayaloid traction ,tractional retinal detachment.

The VMI in patient with DR can influence the emergence ,progression ,and treatment of DR.

The role of posterior hyaloid and vitreous on viteromacular interface abnormalities The anomalous separation of vitreous cortex from ILM can lead to abnormal vitreomacular interface. This separation can happen when liquefaction occur faster than detachment of the vitreous cortex or when an abnormal adhesion of the vitreous cortex to the ILM occur.

The VMI abnormalities in DR include I. Vitreomacular adhesion The International Vitreomacular Traction Study group has defined the vitremacular adhesion as specific stage of vitreous separation when partial detachment of the vitreous in perifoveal area has occurred without any abnormalities to the retinal contour.

II. Vitreomacular traction There is abnormal vitreous adhesion, there can be excessive traction on the macula from the vitreous that change the contour of foveal surface. By OCT any distortion of foveal contour together with partial posterior vitreous detachment is considered vitreomacular traction . In accordance with the International Vitreomacular Traction Study Group definition vitreomacular traction can be classified as focal or broad based on horizontal area of adhesion.

III. Cystoid macular edema The vitreous has been implicated as a cause of macular edema via mechanical and physiologic mechanisms.One of the most constructive hypothesis on how vitreomacular traction may result in macular edema was given by Schubert in 1989,and was summarized by Bringmann and Wiedmann Vitro retinal traction can also exert forces at the level of retinal pigment epithelium ,which can eventually result in morphological retinal pigment epithelial changes .

IV. Epiretinal membrane The epiretinal membrane is a cellular proliferation that creates a semi translucent, fibrocellular proliferation on the surface of the inner retina. Because epiretinal membrane contain contractile cellular elements they can be associated with retinal folding and macular thickening thereby leading to decreased visual acuity, metamorphopsia, monocular diplopia .

V. Full thickness hole Is a full thickness defect in the fovea, include the complete interruption of all retinal layers from the ILM to the retinal pigment epithelium. antero posterior traction, secondary to abnormal attachment at the fovea, and tangential contraction of the perifoveal vitreous cortex may be responsible for the development of the macular hole.

VI. Lamellar holes These include an irregular foveal contour, a defect or break in the inner fovea, a splitting of the inner and outer retina , lack of a full thickness foveal defect, and intact photo receptors.

VII. Macular pseudo hole By OCT the pseudo hole has no loss of retinal tissue. They have invaginated or heaped foveal edge, an epiretinal membrane with a central opening ,and a steep macular contour to the central fovea .the steep foveal contour creates the appearance of hole, even though there is no loss of retinal tissue.

Aim of work Primary outcome : To evaluate the changes in vitreomacular interface in diabetic retinopathy by using Spectral Domain Ocular Coherence Tomography ( SD OCT) Secondary outcome : To evaluate other macular changes in Spectral Domain Ocular Coherence Tomography ( SD OCT) in diabetic patient with vitreomacular interface abnormalities

ELIGIBILITY:
Inclusion Criteria:

* diabetic patient with or without treatment and with or without evidence of vitreomacular traction on clinical examination

Exclusion Criteria:

* diabetic patient with unclear media as dense cataract,
* vitreous Hemorrhage and corneal opacity

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: diabetic male and female patient with age between 12 and 70 years who live in Asiut city
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
measuring visual acuity by snellen chart | two hours
  measuring visual acuity by snellen chart full ophthalmic examination dilating the pupil by mydriatic 1-tropicamide1%drop phenylephrine 2.5%eye drop fundus photography is achived by using TRC 8PLUS TOPCON MEDICAL System,Inc OCT imaging is achived by using Spectral domain OCT (hiedelbrge)

CONTACTS AND LOCATIONS:
Overall Officials: abdalnaser kamil, Study Chair — Asiut university

IPD SHARING:
Plan to Share IPD: Yes
all IPD data will be shared include the age of the patient his heath condition an all information regarding his vision and ophthalmic data and fudus photoes and OCT imaging
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the IPD will be available 2019 and for two years
Access Criteria: the IPD wiil be shared in print out form and C.D form and will be shared with Dr sharaf. mohamed and Dr abdlanaser .Kamil

REFERENCES:
- [Result] 1- Agarwal D, Gelman R, Ponce CP, Stevenson W, and . Christoforidis J B the vitreo macular interface abnormalities in diabetic retinopathy . review. . journal of ophthalmology . 2015. 2- Bottós J, Elizalde J, Arevalo JF, Rodrigues EB, Maia M. Vitreomacular traction syndrome. J Ophthalmic Vis Res 2012 3- Duker JS, Kaiser PK, Binder S, de Smet MD, Gaudric A, Reichel E, et al. The International Vitreomacular Traction Study Group classification of vitreomacular adhesion, traction, and macular hole. Ophthalmology 2013 4- konsantanidis L , Wolfensberger TJ .cystoid macular edema and vitreomacular traction . a review .2015 5- Ryan SJ, Puliafito CA, Davis JL, Parel JM, Milne P. Retina. 4th ed. Philadelphia, PA:Elsevier Mosby; 2006. 6- Chandra A, Charteris DG, Yorston D. Posturing after macular hole surgery: a review. Ophthalmologica 2011
- Available data/document: Study Protocol — https://www.clinicaltrials.gov